CLINICAL TRIAL: NCT07363525
Title: Michigan Initial Experience Using Tigertriever for Thrombectomy
Acronym: MIGHTY
Status: Not yet recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Alex Chebl, Principal Investigator, Henry Ford Health System
Other Study IDs: 18750
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Blood Clot; Thrombectomy; Ischemic Stroke
Keywords: thrombus; Clot; Device; Stroke
MeSH Terms: conditions — Thrombosis; Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Thrombectomy Treated Patients: Patients are enrolled only if the use of the Tigertreiver is used during surgery.
  Interventions: Procedure: Mechanical Thrombectomy

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — You will be asked to provide medical history, take neurological exams in the form of questionnaires, and provide imaging data.

SUMMARY:
The purpose of this research study is to collect data about the effectiveness (i.e. how the device works) and safety (how safe it is to use such a device) of the Tigertriever in restoring blood flow by removing thrombus (or blood clot) from a large intracranial vessel (blood vessel in the brain) in patients experiencing ischemic stroke within 8 hours of symptom onset.

DETAILED DESCRIPTION:
You have been asked to take part in a research study because you have recently been admitted for large vessel occlusion (LVO) and are being treated by Tigertriever.

The treatment is a standard of care (SOC), and if you agree to take part in this study, your participation will include an additional study visit after 3 months. Your study visit will take place at Henry Ford Hospital Neurology or respective collaborator.

For some research studies, such as the one you are being asked to join, it is important that you do not learn the results of certain tests. Whether you intend it or not, sometimes learning this information may make you change your actions and behaviors in ways that could impact the outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with large vessel occlusion (LVO) and treated with the Tigertriever, as per the approved indication.
2. Tigertriever was used as the first line treatment in the target vessel.
3. A signed informed consent.
4. Age ≥ 18.

Exclusion Criteria:

-1. Evidence of acute brain hemorrhage on NCCT or MR at admission. 2. Prior hemorrhage, stroke, thrombolysis, and/or endovascular therapy in the last 3 months.

3. pre-stroke disability (pre-stroke mRS ≥ 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will include male or female subjects age > 18 who present with LVO and are treated with the Tigertriever as per the approved indication.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | From enrollment to 90 days post treatment
  Percentage of participants with a modified Rankin Scale (mRS) score ≤2
Primary Effectiveness Endpoint | By the end of the thrombectomy procdure.
  Percentage of participants with a mTICI Score ≥IIb
Primary Effectiveness Endpoint - mTICI | From time of event to after the first thrombectomy pass.
  Percentage of participants with a mTICI Score ≥IIb after the first pass

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will only be shared and used for publication.